CLINICAL TRIAL: NCT04817410
Title: Emergency Department Initiated Oral Naltrexone for Patients With Moderate to Severe Alcohol Use Disorder: A Pilot Feasibility Study
Brief Title: ED Initiated Oral Naltrexone for AUD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ethan Cowan, Professor of Emergency Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-21-00278
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
Keywords: Medication Assisted Treatment; Emergency Department; Naltrexone
MeSH Terms: conditions — Alcoholism; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Naloxone (Experimental): Oral Naltrexone initiation
  Interventions: Drug: Emergency Department Initiated Oral Naltrexone

INTERVENTIONS:
Drug: Emergency Department Initiated Oral Naltrexone — Emergency Department Initiated Oral Naltrexone

SUMMARY:
This study will recruit Emergency Department (ED) patients with moderate to severe alcohol use disorder (AUD) who are interested in initiating medication assisted treatment (MAT). The study is split into two phases. The first phase (N=10) will use implementation science strategies to strengthen existing non-targeted ED based AUD screening program and optimize feasibility, acceptability, and linkage pathways. The second phase (N=20) will incorporate lessons learned from phase 1 to initiate ED patients on MAT for AUD in the form of oral naltrexone. The primary outcome for both phase 1 and phase 2 is engagement in comprehensive addiction treatment at 14 and 30 days post enrollment.

DETAILED DESCRIPTION:
Overview

The study will be comprised of two components outlined below:

1. Site Implementation Component

   In this component implementation science strategies will be used to strengthen existing non-targeted ED based AUD screening program and optimize feasibility, acceptability and linkage pathways. Three specific aims are to, 1) optimize registered nurse (RN) driven non-targeted alcohol use screening supplemented with secondary screening using DSM-5 criteria for AUD and an SBIRT (screening, brief intervention and referral to treatment) intervention administered by trained staff. 2) During a 3-month period, use continuous quality improvement methods to decrease the time for completion of AUD screening to an interval that is acceptable to ED patients and ED providers and 3) Assess willingness to initiate oral naltrexone among ED patients with moderate to severe AUD. Ten (10) patients will be enrolled in phase 1.
2. Oral Naltrexone Feasibility Component

In this component the study team aims to assess the feasibility of initiating treatment in ED patients with moderate to severe AUD on oral naltrexone, an evidence based and accepted standard of care treatment for AUD. Specifically, 1) over an 8-month period the study team aims to identify 20 patients with moderate to severe AUD eligible and interested in immediate initiation of oral naltrexone. Consenting patients will be receive a standard SBIRT intervention and be provided with immediate oral naltrexone initiation in the ED with a 14-day starter pack at the time of ED discharge. All participants will receive facilitated linkage to comprehensive out-patient care. 2) The study team aims will evaluate the impact of immediate ED initiated oral naltrexone with the primary outcome being engagement in comprehensive addiction care at 14 and 30 days post enrollment. Secondary outcomes include medication adherence, changes in daily alcohol consumption, number of heavy drinking days, hospital admissions and ED utilization, transition to long-acting injectable naltrexone and alcohol craving. 3) Lastly, the study team will collect data on recruitment and attrition rates, as well as means and standard deviations for key measures that will be needed to plan a definitive randomized controlled trial of ED-initiated oral naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients 18 years of age or older
* Treated in the ED during screening hours
* Moderate to severe AUD as determined by DSM-5 criteria
* Able to speak and understand English
* Medically stable for an interview as determined by their primary ED provider
* Willing and able to consent to study participation
* Two points of contact available for follow-up

Exclusion Criteria:

* ED patients younger than 18 years of age
* Medically or psychiatrically unstable as determined by the ED provider
* Unable to speak or understand English
* Unable to provide consent for study participation
* Past year opioid dependence
* Urine drug screen positive for opioids
* Current or anticipated need for opioid medications for pain
* Anticipated surgical procedure within 14-day of ED visit
* Serologic evidence of liver disease (LFTs 3X normal) within 7 days of enrollment
* Cirrhosis either by PMH or self-report
* Pregnant or breastfeeding
* Lacking contact information for follow-up
* Requiring in-patient admission for medical or psychiatric reasons
* Patient receiving a sexual assault forensics exam (SAFE)
* Patient suspected of having COVID-19
* Patient is actively suicidal or homicidal
* Previously enrolled in either the implementation or feasibility phase of the study
* Be a prisoner or in police custody at the time of the index ED visit
* Be currently (anytime within the last 14 days) enrolled in formal addiction treatment, including by court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Cowan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective single-arm, open-label, nonrandomized clinical trial in patients with moderate to severe AUD presenting to the Mount Sinai Beth Israel ED between September 2021 and October 2023.
Period: Overall Study
Arm/Group | Oral Naloxone
Started | 29
Completed | 21
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Oral Naltrexone: Oral Naltrexone
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [30 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 21
Highest Level of Education [Count of Participants; unit: Participants]
  Some high school, no diploma | 4
  high school graduate/GED equivalent | 3
  Technical/trade/vocational school | 2
  Junior (2 year) college | 1
  Some college (4 year college or university) | 5
  College graduate (4 year college or university) | 3
  Post-college/graduate degree | 1
  Missing | 2
Estimated Total Income [Count of Participants; unit: Participants]
  Less than $1,00 | 2
  $10,001-$20,00 | 1
  20,001-$40,000 | 3
  $40,001 or more | 8
  Don't know/missing | 7
Past-year Employment Status [Count of Participants; unit: Participants]
  Unemployed | 4
  Employed | 7
  Disabled, permanently or temporarily | 3
  Other | 7
Health Insurance Coverage [Count of Participants; unit: Participants]
  Covered by health plan | 18
  Not Covered by health plan | 3
Concerned about stable housing over the next two months [Count of Participants; unit: Participants]
  Yes | 9
  No | 12
Incarcerated in the last 12 months [Count of Participants; unit: Participants]
  Yes | 0
  No | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled and Receiving Formal Addiction Treatment at Day 14
Description: Number of participant enrolled with engagement in care of comprehensive addiction treatment
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Groups:
- Oral Naltrexone: Received at least one dose of oral naltrexone
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
Participants
  Engaged in treatment at 14-days | 6
  Not engaged in treatment at 14-days | 15

2. Primary Outcome: Number of Participants Enrolled and Receiving Formal Addiction Treatment at Day 30
Description: Number of participant enrolled with engagement in care of comprehensive addiction treatment
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Participant Characteristics: Received at least 1 dose of oral naltrexone
Arm/Group | Enrolled Participant Characteristics
Number analyzed (Participants) | 21
Participants
  Engaged in treatment at 30-days | 7
  Not engaged in treatment at 30-days | 14

3. Secondary Outcome: Number of Alcoholic Drinks Per Day
Description: Baseline
Time Frame: 7-days prior to enrollment to day of enrollment (baseline)
Measure: Median (Inter-Quartile Range); unit: # of drinks consumed per day
Groups:
- Oral Naltrexone: Received at least 1 dose of oral naltrexone
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
# of drinks consumed per day | 4.29 [2.29 to 7.57]

4. Secondary Outcome: Number of Daily Drinks
Description: 30-days
Time Frame: 30-days
Population: 30-days
Measure: Median (Inter-Quartile Range); unit: # of drinks consumed per day
Arm/Group | Enrolled Participant Characteristics
Number analyzed (Participants) | 21
# of drinks consumed per day | 0.73 [0 to 2.81]

5. Secondary Outcome: Daily Alcohol Craving Scale
Description: Daily alcohol craving scale using Qualtrics - Full scale from 0 to 36, higher score represents more severity.
Time Frame: up to 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enrolled Participant Characteristics
Number analyzed (Participants) | 21
score on a scale | 8.27 [4.65 to 11.75]

6. Secondary Outcome: Guidelines Regimen Information Program (GRIP) Guide at Day 14
Description: Adherence to daily oral naltrexone measured using Guidelines Regimen Information Program (GRIP) guide - GRIP guide is a self-report to assess adherence, with 6 categorical items: excellent, very good, good, fair, poor, and very poor. The maximum value is 6 and the minimum value is 1. Higher scores mean better adherence.
Time Frame: Day 14
Population: Adherence to daily oral naltrexone measured using Guidelines Regimen Information Program (GRIP) guide - GRIP guide is a self-report to assess adherence, with 6 categorical items: excellent, very good, good, fair, poor, and very poor. The maximum value is 6 and the minimum value is 1. Higher scores mean better adherence.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
units on a scale | 4.5 [3 to 5]

7. Secondary Outcome: Guidelines Regimen Information Program (GRIP) Guide at Day 30
Description: Adherence to daily oral naltrexone measured using the Guidelines Regimen Information Program (GRIP) guide - GRIP guide is a self-report to assess adherence, with 6 categorical items: excellent, very good, good, fair, poor, and very poor. The maximum value is 6 and the minimum value is 1. Higher scores represent better adherence.
Time Frame: Day 30
Population: Adherence to daily oral naltrexone measured using the Guidelines Regimen Information Program (GRIP) guide - GRIP guide is a self-report to assess adherence, with 6 categorical items: excellent, very good, good, fair, poor, and very poor. The maximum value is 6 and the minimum value is 1. Higher scores represent better adherence.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
units on a scale | 4 [4 to 5]

8. Secondary Outcome: Number of Pills in Bottle at Day 14
Description: Adherence to daily oral naltrexone measured using pill counts.
Time Frame: Day 14
Population: Pill count at day 14. Note: Participants did not return to clinic so pill counts were not collected.
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Pills in Bottle at Day 30
Description: Adherence to daily oral naltrexone measured using pill counts.
Time Frame: Day 30
Population: Pill counts at day 30 Note: Participants did not return to clinic so pill counts were not collected.
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Heavy Drinking Days
Description: Number of heavy drinking days defined as 4 or more drinks for a woman or 5 or more drinks for a man on the same occasion in a 24 hour period.
Time Frame: up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
days | 0.0 [0 to 0.17]

11. Secondary Outcome: Health Services Utilization Survey
Description: Participants indicated the number of inpatient admissions, outpatient visits and emergency department visits over the preceding 7-days at baseline up to 30-days. Comparison of total reported admissions or visits were made using the Friedman test. No admissions or visits counted as a 0 for comparing across timepoints. If no response was provided at any of the three time points, the participant data was not used in the comparison.
Time Frame: up to 30-days
Population: Participants indicated the number of inpatient admissions, outpatient visits and emergency department visits over the preceding 7-days at baseline, 14-days and 30-days. Comparison of total reported admissions or visits were made using the Friedman test. No admissions or visits counted as a 0 for comparing across timepoints. If no response was provided at any of the three time points, the participant data was not used in the comparison.
Measure: Median (Inter-Quartile Range); unit: number of occurrences
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
number of occurrences
  Inpatient Admissions - baseline | 0 [0 to 0]
  outpatient visits -baseline | 0 [0 to 1]
  ED visits - baseline | 0 [0 to 0]
  Inpatient admissions-day 14 preceding 7-days at baseline) | 0 [0 to 0]
  Outpatient visits-day 14 | 0.5 [0 to 1]
  Emergency Department Visits - day 14 | 0 [0 to 0]
  Inpatient admission - day 30 | 0 [0 to 0]
  Outpatient visits - day 30 | 0 [0 to 1]
  ED visits - day 30 | 0 [0 to 0]

12. Secondary Outcome: Number of Unhealthy Days Assessed by Health Related Quality of Life (HRQoL)
Description: Number of unhealthy days using the HRQoL. The HRQoL assesses core health days and activity limitations. Self-reported general health was collected on a 5-item scale ranging from: excellent, very good, good, fair, and poor. An unhealthy days score was obtained by summing the number of physically unhealthy and mentally unhealthy days. The minimum score is 0 and the maximum score is 30 unhealthy days, even if the number of unhealthy days totals more than 30. If no response was provided at the time points under comparison, the participant data was not used in the comparison.
Time Frame: Day 30
Population: Self-reported general health was collected on a 5-item scale ranging from: excellent, very good, good, fair, and poor. An unhealthy days score was obtained by summing the number of physically unhealthy and mentally unhealthy days. The minimum score is 0 and the maximum score is 30 unhealthy days.
Measure: Median (Inter-Quartile Range); unit: unhealthy days
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 18
unhealthy days | 11.5 [0 to 30]

13. Secondary Outcome: The Patient Rated Inventory of Side Effects (PRISE) Survey
Description: Medication side effects of oral naltrexone measured using PRISE survey - is a patient self-report measure used to identify and evaluate the tolerability of side effect symptom. This scale is a 7-item assessment of the side effects in the following symptom areas; gastrointestinal, heart, skin, nervous system, eyes/ears, genital/urinary, sleep, sexual functioning, and other. Each domain has multiple symptoms and for each domain the patient rates whether these symptoms are tolerable or distressing. Higher score represents more side-effects. What is reported below are the number of participants reporting side effects for each symptom.
Time Frame: Day 30
Measure: Number; unit: participants
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
participants
  Gastrointestinal | 10
  Heart | 6
  Skin | 3
  Nervous System | 6
  Genital/Urinary | 8
  Sleep | 10
  Sexual Functioning | 6
  Other | 11
  Eyes/Ears | 4

14. Secondary Outcome: AUD Program Satisfaction Survey at Baseline
Description: Three elements of satisfaction were assessed: 1) convenience of screening, 2) difficulty of screening and 3) satisfaction with screening. Each question could be scored on scale of 0-6. For convenience of screening, lower numbers indicated more convenience. For difficulty of screening, lower numbers represent less difficulty. For satisfaction, higher numbers represent greater satisfaction.
Time Frame: Baseline
Population: Three elements of satisfaction were assessed: 1) convenience of screening, 2) difficulty of screening and 3) satisfaction with screening. Each question could be scored on scale of 0-6. For convenience of screening, lower numbers indicated more convenience. For difficulty of screening, lower numbers represent less difficulty. For satisfaction, higher numbers represent greater satisfaction.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Naltrexone
Number analyzed (Participants) | 21
Participants
  Satisfaction with screening: 0 | 1
  Satisfaction with screening: 1 | 1
  Satisfaction with screening: 2 | 1
  Satisfaction with screening: 3 | 0
  Satisfaction with screening: 4 | 1
  Satisfaction with screening: 5 | 1
  Satisfaction with screening: 6 | 16
  Convenience of screening: 0 | 14
  Convenience of screening: 1 | 1
  Convenience of screening: 2 | 1
  Convenience of screening: 3 | 2
  Convenience of screening: 4 | 0
  Convenience of screening: 5 | 1
  Convenience of screening: 6 | 2
  Difficulty of screening: 0 | 13
  Difficulty of screening: 1 | 3
  Difficulty of screening: 2 | 2
  Difficulty of screening: 3 | 0
  Difficulty of screening: 4 | 0
  Difficulty of screening: 5 | 1
  Difficulty of screening: 6 | 2

15. Secondary Outcome: Number of Participants Who Transition to LA Injectable
Description: Number of participants who transition from oral to long acting injectable naloxone.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participant Characteristics
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 30-days
Arm/Group | Oral Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Due to the nonrandomized design, lack of a nontreatment control and small sample size, drawing inferences about efficacy of ED-initiated naltrexone on short-term engagement in care is not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04817410/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT04817410/ICF_001.pdf